CLINICAL TRIAL: NCT03804112
Title: TransIent Perivascular Inflammation of the Carotid Artery (TIPIC) Syndrome: Clinical and Radiological Follow-up
Acronym: TIPIC-UNV
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: MOA_2018_2
Record Dates: First submitted 2019-01-11; First posted 2019-01-15 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Cervical Pain; Vasculitis
MeSH Terms: conditions — Neck Pain; Vasculitis | interventions — Echocardiography, Doppler; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Ultrasound exam with Doppler — Ultrasound exam of the neck to search a perivascular inflammation at the level of the carotid bifurcation.
Biological: Blood samples — blood count , CRP and viral serologies (herpes virus, chlamydia, mycoplasma),

SUMMARY:
TIPIC syndrome (previously called carotidynia) is a rare entity of unknown cause, where the patient has a temporary cervical pain associated with a suggestive inflammation around the carotid artery. Usually considered as a unique and benign episode, some patients have recurrences and the follow-up is usually short. In this study the investigators aim to evaluate patients who presented a TIPIC episode at least 3 months before, clinically and with a cervical doppler ultrasound

ELIGIBILITY:
Inclusion Criteria:

- Patients with at least one episode of TIPIC syndrome for more than 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patient previously identified with a TIPC syndrom
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2018-12-17 (Actual); Primary Completion 2020-02-18 (Actual); Study Completion 2020-02-18 (Actual)

PRIMARY OUTCOMES:
Assess the incidence of recurrence of TIPIC syndrome after a first episode | 1 year

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - CHU de Montpellier, Montpellier
  - Hôpital Pitié Salpêtrière, Paris
  - Centre Hospitalier de Saint-Anne, Paris
  - Fondation Ophtalmologique A. de Rothschild, Paris
  - CHU de Toulouse, Toulouse
  - CHU de TOURS, Tours

REFERENCES:
- [Derived] Obadia M, Nasr N, Volle G, Charbonneau F, Guillaume J, Naggara O, Sadik JC, Lecler A. Long-term clinical and ultrasound follow-up after transient perivascular inflammation of the carotid artery (TIPIC) syndrome: a multicenter study. Cephalalgia. 2024 Feb;44(2):3331024241230247. doi: 10.1177/03331024241230247. PMID 38318645